CLINICAL TRIAL: NCT02653859
Title: Evaluate the Auxiliary Diagnostic Value of Circulating Tumor Cells(CTC) in Benign and Malignant Lung Nodules
Brief Title: Evaluate the Auxiliary Diagnostic Value of Circulating Tumor Cells in Benign and Malignant Lung Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GenoSaber (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC2015-02
Record Dates: First submitted 2016-01-03; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-10

CONDITIONS: Solitary Pulmonary Nodule
Keywords: CTC; PCR
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
By testing the CTC number of new solitary pulmonary nodule patient, evaluating the correlation of CTC number and benign and malignant lung nodules auxiliary diagnosis, the correlation of CTC number and the size of lung nodules of the malignant patients, the correlation between the CTC number and subtypes of malignant lung nodules patients.The CTC and tumor markers will be detected before the patient received treatment. Tumor markers include Pro-GRP, NSE, CEA, CYFRA211, SCC.

ELIGIBILITY:
Inclusion Criteria:

* New Solitary Pulmonary Nodule patients
* first visit patient
* Heart, liver and kidney function is normal.
* 18-80 years old.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Blood collection time is not in the scheduled time.
* The plasma sample hemolysis or condensation.
* Whole blood samples less than 3 ml.
* poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New Solitary Pulmonary Nodule
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The number of circulating tumor cells will be detected in baseline by Immunomagnetic negative screening and targeted polymerase chain reaction(PCR) method. | 1 months
  The 3 mL of blood will be taked with each patient for CTCs detection.

SECONDARY OUTCOMES:
The concentration of the tumor marker of pro gastrin releasing peptide(Pro-GRP) will be detected in baseline by Electrochemical luminescence. | 1 months
  The 2 mL of serum will be extracted.
The concentration of the tumor marker of neurone specific enolase(NSE) will be detected in baseline by Electrochemical luminescence. | 1 months
  The 2 mL of serum will be extracted.
The concentration of the tumor marker of carcinoembryonic antigen(CEA) will be detected in baseline by Electrochemical luminescence. | 1 months
  The 2 mL of serum will be extracted.
The concentration of the tumor marker of cytokeratin 19 fragments(CYFRA211) will be detected in baseline by Electrochemical luminescence. | 1 months
  The 2 mL of serum will be extracted.
The concentration of the tumor marker of squamous cell carcinoma antigen(SCC) will be detected in baseline by Electrochemical luminescence. | 1 months
  The 2 mL of serum will be extracted.